CLINICAL TRIAL: NCT06771297
Title: The Effect of Education Given to Patients Undergoing Rhinoplasty Surgery on Involuntary Thoughts and Recovery Quality
Brief Title: Education's Impact on Involuntary Thoughts and Healing in Rhinoplasty Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Turgut Sohret, PhD student, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AtaturkUniNursing
Record Dates: First submitted 2024-06-26; First posted 2025-01-13 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Rhinoplasty; Nursing Education
Keywords: rhinoplasty; nursing; involuntary thought; quality of recovery; education
MeSH Terms: interventions — Nursing Education Research

STUDY DESIGN:
Intervention Model Description: The population of the research is Iğdır, Dr. Patients who underwent rhinoplasty surgery and applied to Nevruz Erez State Hospital Plastic Surgery Clinic and Ear, Nose and Throat Clinic between January 2024 and December 2024 were included. The sample will consist of 82 patients selected by simple random sampling method and meeting the research criteria. The sample was determined by G-Power.
Who Masked: Participant
Masking Description: Patients were not told which group they were in. In this way, single blinding was achieved.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care and nursing education (Experimental): Nursing training will be provided the day before the surgery.
  Interventions: Other: nursing education
- standard care (Other): Nursing training will not be provided and will only receive standard care in the hospital.
  Interventions: Other: nursing education

INTERVENTIONS:
Other: nursing education — Nursing training will be given before rhinoplasty surgery. As a result, patients' involuntary thoughts and quality of recovery will be questioned.

SUMMARY:
With planned trainings prepared by taking into account the needs of patients and given by nurses, levels of anxiety and involuntary thoughts can be reduced and the quality of service and recovery can be increased. In this context, this research was planned to determine the effect of preoperative education given to patients undergoing rhinoplasty surgery on involuntary thoughts and recovery quality.

DETAILED DESCRIPTION:
Rhinoplasty , nose shape And function disorders elimination for the purpose of often applied surgical One is the procedure . Higher ego respect , aesthetics your concerns elimination And life of the quality increasing for the purpose of today rhinoplasty And other aesthetic surgical of procedures APPLICATION in frequency increase surgery while being observed to the process connected aspect developing anxiety because of dissatisfaction And pain like negative seeing the experiences frequency increasing . Age , personal features , history experiences And to do to applications connected aspect individual Differences by showing together hospital lying down require , general anesthesia under implementation , specific One duration work vital And social from life far to stay like A lot factor rhinoplasty surgery before And after that individuals anxiety to live From where is happening . Moreover surgical of the procedure aesthetic for purposes being done to have surgery after that get will be conclusion with relating to obscurity sense of And external appearances given high importance patients anxiety levels affecting other factors aspect is shown . To do to transactions aimed at information lack of patients anxiety level affecting -most basis from factors someone is is stated . patients requirements into consideration by taking prepared And nurses by given planned trainings with anxiety And request female thought levels reducing And patients improvement of the quality increasing is intended .

patients requirements into consideration by taking prepared And nurses by given planned trainings with anxiety And request female thought levels can be reduced And service And improvement of the quality can be increased . In this context This research rhinoplasty surgery will be to patients operation pre- given your education request female thoughts And improvement to the quality effect to determine for the purpose of was the plan .

Approach and Methods to be Applied:

of research Place and Time of Making : This research was conducted by Iğdır Dr. It will be carried out at Nevruz Erez State Hospital, Plastic Surgery Clinic between January 2024 and December 2024.

Population and Sample of the Research: Population of the research, Iğdır Dr. Nevruz Erez State Hospital, Plastic Surgery Clinic Patients who underwent rhinoplasty surgery and applied between January 2024 and December 2024 will be created. The sample will consist of 82 patients selected by simple random sampling method and meeting the research criteria.

Method of the research : It was planned as a randomized controlled experimental.

of research Variables : Dependant Variables : Prompt Female Thoughts Scale , Surgery Post Improvement index Independent Variables : surgery pre- education Control Variables : Patient's age , gender , marital status , education level , more before operation being situation , else One health problem being status Data Collection and Initiatives: Research for First of all , Ataturk University Medicine Faculty Ethic From the Board approval And of research will be carried out from hospitals written permissions will be taken . Necessary permissions after receiving After , January 2024- December 2024 between Iğdır Dr. Research at Nevruz Erez State Hospital, Plastic Surgery Clinic to join acceptance who makes And sample being elected to the criteria wake up patients to work including will be . Research of your data "Patient Introduction " in the meeting Form ", " Request Female Thoughts Scale " and " Surgery Post Improvement Index " will be used . Data collecting tools This way Will be implemented : Researcher by surveys face to the face meeting technique using to patients will be filled . Control in the group patients , surgery One day Before Patient Introduction form And Request Female Thoughts scale will be implemented . Operation in the morning Request Female Thoughts scale again will be implemented . Operation post- whereas discharged while being And discharged 1 week after later Operation Post Improvement index will be applied. Patients in the control group will receive routine nursing care.

the experimental group to patients from surgery One day Before Patient Introduction form And Request Female Thoughts scale will be implemented . Later computer in the environment prepared slide with his offering rhinoplasty process pre- And may develop after complications And at home care process with relating to education will be given . Later prepared education booklet to patients will be given . Operation in the morning Request Female Thoughts scale again will be implemented . Operation post- whereas discharged while being And discharged 1 week after later Operation Post Improvement index will be applied.

Data Collection Tools:

Introductory Information Form: It consists of questions containing the demographic characteristics of the patient, prepared by the researchers in line with the literature for the purpose of collecting research data.

Operation Pre Request Female Thoughts scale Operation pre- in patients happened anxiety to research And operation pre- of anxiety fast One way evaluation to ensure For this purpose, Crockett et al. by has developed . of scale Turkish validity And reliability Cakir and by Karabulut has been made . Control loss concern size And process until later related anxiety size to be about into two subdimensions has . out of 20 items formed This each question of the scale for evaluation: (0) never , (1) sometimes , (2) often chic and (3) mostly shaped and 4-point Likert to type has . From scale 0-60 point can be obtained . 15 or more high One score , clinic aspect important to anxiety reaching patients Trustworthy One way detection it does .

Postoperative Recovery Index (PRI): The Postoperative Recovery Index was developed by Butler et al. in 2012 (26) and was validated in Turkish by Cengiz and Aygin (2019) (27). The index consists of 5 sub-dimensions and 25 items. The sub-dimensions include psychological symptoms, physical activities, general symptoms, bowel symptoms, and desire-related symptoms. Sub-dimension scores are calculated by summing the relevant item scores and taking their arithmetic mean. The total score is determined by summing all item scores and calculating the arithmetic mean. Higher scores indicate greater difficulties in postoperative recovery, while lower scores suggest easier recovery (27). In the study by Cengiz and Aygin, the Cronbach's alpha coefficient for the PRI was determined to be 0.96 (27).

Evaluation of Data: Statistical Package for the Social Science (SPSS) statistical package will be applied in the coding and statistical analysis of the data. Descriptive statistics, t-test for dependent and independent groups, and correlation tests will be used to evaluate the data.

Ethical Aspect of the Research: In order to conduct the research, Ethics Committee approval will be obtained from Atatürk University Faculty of Medicine Ethics Committee Presidency. In addition, Iğdır Dr. where the research will be carried out . Legal permissions will be obtained from Nevruz Erez State Hospital . Since answers must be given voluntarily in all research that obtains information, importance will be given to the voluntary participation of individuals to be included in the research. In addition, their approval (principle of informed consent) will be obtained verbally after the purpose of the research and the purposes for which the results will be used are explained. The "Respect for Autonomy" principle will be fulfilled by stating that they are free to participate in the research or not, and the "Confidentiality and Protection of Confidentiality" principle will be fulfilled by informing the patients participating in the research that their information will be kept confidential. Since individual rights must be protected in research, the Declaration of Helsinki on human rights will be adhered to during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Experienced planned nose surgery for the first time,
2. Volunteer to participate in the research,
3. 18 years and above,
4. Mental status is healthy,
5. Having no vision, hearing or speech problems,
6. Patients who speak Turkish will be included in the study.

Exclusion Criteria

1. Having had nose surgery before,
2. Communication is a problem,
3. Patients who do not want to participate in the study voluntarily will not be included.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Preoperative Intrusive Thoughts Inventory (PITI) | surgery day morning (1 day)
  This scale aims to investigate preoperative anxiety in patients and provide a rapid assessment of this anxiety. It consists of two sub-dimensions: concern about loss of control and concern related to post-procedural outcomes. The scale contains 20 items, with responses evaluated on a 4-point Likert scale ranging from (0) never, (1) sometimes, (2) often, to (3) mostly. Scores range from 0 to 60, with a score of 15 or higher reliably identifying patients with clinically significant anxiety.
Preoperative Intrusive Thoughts Inventory (PITI) | Day before surgery (1 day)
  This scale aims to investigate preoperative anxiety in patients and provide a rapid assessment of this anxiety. It consists of two sub-dimensions: concern about loss of control and concern related to post-procedural outcomes. The scale contains 20 items, with responses evaluated on a 4-point Likert scale ranging from (0) never, (1) sometimes, (2) often, to (3) mostly. Scores range from 0 to 60, with a score of 15 or higher reliably identifying patients with clinically significant anxiety.
  Time Frame: 1 day

SECONDARY OUTCOMES:
Postoperative Recovery Index (PRI) | 1st day after surgery
  The index consists of five sub-dimensions: psychological symptoms, physical activities, general symptoms, bowel symptoms, and desire-related symptoms. Scores range from 25 to 125. The total score for the PRI general survey is calculated by summing all 25 items and taking the arithmetic mean. Higher scores indicate greater difficulties in postoperative recovery, while lower scores suggest an easier recovery process.
Postoperative Recovery Index (PRI) | 1st week after surgery
  The index consists of five sub-dimensions: psychological symptoms, physical activities, general symptoms, bowel symptoms, and desire-related symptoms. Scores range from 25 to 125. The total score for the PRI general survey is calculated by summing all 25 items and taking the arithmetic mean. Higher scores indicate greater difficulties in postoperative recovery, while lower scores suggest an easier recovery process.
  Time Frame: 1 day and 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Neziha Karabulut, Prof.Dr., Study Chair — Researcher; Turgut Şöhret, Lecturer, Study Chair — Researcher; Yasemin Ay Karadaş, Lecturer, Study Chair — Researcher
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: January 2024- December 2024

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/17567344/
- See also: Related Info — https://www.longdom.org/open-access-pdfs/development-and-validation-of-the-post-operative-recovery-index-for-measuring-quality-of-recovery-after-surgery-2155-6148.1000267.pdf